CLINICAL TRIAL: NCT05346172
Title: The Clareon PanOptix Trifocal IOL: A Study of Patient Satisfaction and Visual Performance
Brief Title: The Clareon PanOptix Trifocal IOL: Visual Outcomes and Patient Satisfaction
Status: Completed | Type: Observational
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2111 Clareon PanOptix
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: PanOptix or PanOptix Toric IOL — Patients who previously underwent cataract surgery with the PanOptix or PanOptix Toric IOL in both eyes.

SUMMARY:
This will be a single arm, open-label, prospective study of patient-reported outcomes of patients with bilateral implantation of the Panoptix or Panoptix Toric implant.

DETAILED DESCRIPTION:
The PanOptix trifocal lens by Alcon was introduced in 2015 and is currently in use in over 70 countries. Its outcomes on the AcrySof platform are well documented and highly appealing to patients and clinicians.,, Clinicians no longer need to routinely target monovision or modified monovision to provide a range of vision. With the release of the Clareon material for this lens, questions remain about how the new lens material will influence patient satisfaction and uncorrected visual performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataract and otherwise healthy eyes, not exhibiting any significant ocular morbidity that would be expected to influence outcome measures.
* Patients implanted with Clareon PanOptix or Clareon Panoptix Toric lenses bilaterally within 6 months of the survey administration.

Exclusion Criteria:

* Patients with visually significant comorbidities (corneal, retina, optic nerve disease) that could affect their satisfaction with surgery
* Patients with surgical complications either during or after surgery (capsule tears, iris trauma, decentered IOL, cystoid macular edema, etc.)
* Patients with previous refractive surgery within the past 6 months prior to cataract surgery
* Patients with > grade 1 posterior capsule opacity at their last visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reporting "not at all" or "just a little" when asked, "With or without glasses, how much do you notice glare or haloes around lights in dim light situations?" | Up to 6 months
  Percentage of patients who notice glare or haloes around lights in dim light situations

SECONDARY OUTCOMES:
Percentage of postoperative patients who report "rarely" when asked "How often do you need glasses to see the computer?" | Up to 6 months
  How often do you need glasses to see the computer.
Percentage of postop patients who report they do not require reading glasses for various activities when asked "For what types of activities do you need glasses to see (other than sunglasses)?" | Up to 6 months
  Percentage of postoperative patients who report that they do not require glasses for varous activities.

OTHER OUTCOMES:
Percentage of patients reporting "very satisfied" when asked, "Overall, how satisfied are you with your vision after your latest surgery?" | Up to 6 months
  Percentage of patients satisfied with their vision after surgery
Percentage of patients who report "very satisfied" or " Somewhat satisfied" to the same question. | Up to 6 months
  Percentage of patients who report "very satisfied" or " Somewhat satisfied" to the same question.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Harvard Eye Associates, Laguna Hills, California
  - Florida Vision Institute, Stuart, Florida
  - IllinEye Consulting, Evansville, Illinois